CLINICAL TRIAL: NCT00039988
Title: Treatment of Multiple Sclerosis With Copaxone (Glatiramer Acetate) and Albuterol
Brief Title: Treatment of Multiple Sclerosis With Copaxone and Albuterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT AMS01; ACE Study AMS01
Record Dates: First submitted 2002-06-18; First posted 2002-06-20 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Autoimmune Diseases; Multiple Sclerosis
Keywords: Treatment Outcome; Multiple Sclerosis; Albuterol; Copolymer 1
MeSH Terms: conditions — Autoimmune Diseases; Multiple Sclerosis | interventions — Glatiramer Acetate; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Experimental): Participants will receive Copaxone and albuterol placebo
  Interventions: Drug: Glatiramer acetate; Drug: Albuterol placebo
- 2 (Experimental): Participants will receive Copaxone and albuterol
  Interventions: Drug: Glatiramer acetate; Drug: Albuterol

INTERVENTIONS:
Drug: Glatiramer acetate — 20 mg administered subcutaneously daily
Drug: Albuterol — 2 mg or 4 mg oral capsules taken daily
  Arms: 2
Drug: Albuterol placebo — Oral placebo capsules will be taken daily
  Arms: 1

SUMMARY:
The purpose of this study is to determine the effects of glatiramer acetate (Copaxone) alone compared to Copaxone plus albuterol in patients with Multiple Sclerosis (MS).

MS is thought to be an autoimmune disease of the central nervous system. Certain white blood cells of the immune system become abnormally active and mistakenly attack the myelin of nerve fibers. Myelin is a fatty sheath that surrounds nerve fibers and insulates the nerve like insulation around an electrical wire. Without proper myelin insulation, messages sent between the brain and other parts of the body may be confused or fail completely. Damage to myelin causes the symptoms of MS. The most common form of MS is known as relapsing-remitting (RR), where partial or total recovery occurs after attacks. Four therapies are currently approved for the treatment of MS. These therapies, however, are only moderately effective and can cause undesirable side effects. For this reason, there is a need to find new therapies that have minimal side effects and may stop the disease from getting worse.

DETAILED DESCRIPTION:
MS is a chronic inflammatory disease of the central nervous system characterized by focal T cell and macrophage infiltrates that lead to demyelination and loss of neurologic function. Four therapies are currently approved for the treatment of MS. Three of these are approved for the treatment of patients with the relapsing-remitting (RR) form of MS, in which patients have clinical exacerbations followed by partial or complete recovery of function. These treatments are only modestly effective and are associated with significant toxicity, often causing patients to delay therapy for significant lengths of time. Thus, there is a need to find therapies with low toxicities that can be administered early during the disease course with the potential for arresting the disease.

During the pre-treatment phase, patients undergo neurological exams, including the extended disability status scale (EDSS), Ambulation Index (AI), disease steps (DS) scale MS functional composite score, PASAT, 9 hole peg test, and the 25 foot walking time. A 12-lead electrocardiogram (EKG) and chest x-ray are performed. Serum chemistry is assessed as well as electrolyte and thyroid stimulating hormone (TSH) levels. A brain MRI (with and without gadolinium), urinalysis, and urine pregnancy test (for women of reproductive potential) are performed. Blood is collected for mechanistic studies. In the treatment phase, patients are assigned randomly to 1 of 2 study arms:

Arm 1: Copaxone plus placebo. Arm 2: Copaxone plus albuterol. At the treatment visits, blood is collected and neurological exams and a brain MRI are performed. A pregnancy test is administered to women of reproductive potential. Neurological exams are performed every 6 months. MRIs are performed at baseline, Year 1, and Year 2. At the end of the study, patients have a complete physical exam, a neurological exam, and a brain MRI.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Have been diagnosed with RR-MS, within 2 years of diagnosis.
* Are 18-55 years old.
* Have RR-MS with evidence of demyelination on MRI scanning of the brain.
* Have extended disability status scale (EDSS) scores between 0 and 3.5.
* Have not taken Copaxone or oral myelin.
* Have not had immunomodulating therapy for the past 3 months.
* Have not taken immunosuppressants.
* Have not had steroid treatment 1 month before entry.
* Have no evidence of active infection or cancer.

Exclusion Criteria

Patients may not be eligible for this study if they:

* Have a normal brain MRI.
* Are not willing to practice contraception (applies to women who are able to have children).
* Are pregnant or breast-feeding.
* Are currently taking any of the following drugs: beta2-adrenergic agonist or antagonist, diuretics, tricyclic antidepressants, or monoamine oxidase inhibitors.
* Have heart, blood, liver, or kidney problems.
* Have a disease that affects blood clotting or lung function.
* Have abnormalities that relate to the endocrine system.
* Have a history of alcohol or drug abuse within 6 months of enrollment.
* Have been diagnosed with primary progressive MS, in which the disease slowly worsens without periods of recovery.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2001-11; Primary Completion 2006-03 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change in each participant's disease status, as measured by the Multiple Sclerosis Functional Composite score (MSFC) | Throughout study
Glatiramer acetate-specific cytokine secretion of IL-13 cytokine secretion and IFN-gamma secretion by glatiramer acetate-reactive T-cell lines | At Months 3, 6, and 12

SECONDARY OUTCOMES:
Change in IL-5 secretion in the supernatants of lines stimulated with glatiramer acetate | Throughout study
Change in percentage of IL-12-producing monocytes by intracytoplasmic staining | Throughout study
Time to first exacerbation | Throughout study
Number and severity of exacerbations | Throughout study
MRI evidence as measured by T2 lesion volume, number of enhancing lesions on T1 weighted images, and measurements of atrophy (brain parenchymal fraction, atrophy index) | At study entry and Months 12 and 24
Expanded Disability Status Scale (EDSS), Ambulation Index (AI), and Disease Steps (DS) scores | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Samia Khoury, Principal Investigator — Brigham and Women's Hospital/Harvard Medical School
Locations (1):
- Brigham and Women's Hospital/Harvard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data access including but not limited to participant level data, is available to the public in the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Result] Khoury SJ, Healy BC, Kivisakk P, Viglietta V, Egorova S, Guttmann CR, Wedgwood JF, Hafler DA, Weiner HL, Buckle G, Cook S, Reddy S. A randomized controlled double-masked trial of albuterol add-on therapy in patients with multiple sclerosis. Arch Neurol. 2010 Sep;67(9):1055-61. doi: 10.1001/archneurol.2010.222. PMID 20837847
- Available data/document: Individual Participant Data Set: Study identifier is SDY471 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY471
- Available data/document: Study Protocol: Study identifier is SDY471 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY471
- Available data/document: Study summary, -design, -adverse events, -medications, -demographics, -lab tests, -mechanistic assays, et al.: Study identifier is SDY471 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY471